CLINICAL TRIAL: NCT06459310
Title: A Phase II Exploratory Clinical Study Investigating the Geroprotective Effect of Metformin in Middle-aged and Elderly People
Brief Title: Pilot Study on Evaluating the Geroprotective Effect of Metformin
Acronym: AGE-M
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Xuanwu Hospital, Beijing (Other)
Collaborators: Institute of Zoology, Chinese Academy of Sciences (Other Government); Beijing Institute of Genomics, Chinese Academy of Sciences (Other Government); Merck Serono Co., Ltd., China (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: lijingxw
Record Dates: First submitted 2024-06-03; First posted 2024-06-14 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Metformin; Aging
Keywords: aging intervention; metformin; aging biomarker; multi-omics; middle-aged and elderly people; molecular clocks; biological age
MeSH Terms: interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Metformin hydrochloride (Experimental): 1000 mg/day Metformin hydrochloride extended-release tablets
  Interventions: Drug: Metformin Hydrochloride tablet
- Placebo group (Placebo Comparator): 1000 mg/day placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Metformin Hydrochloride tablet — Extended release oral tablets, 1000 mg/day, single dose
  Other Names: Metformin
  Arms: Metformin hydrochloride
Drug: Placebo — Oral tablets, 1000 mg/day, single dose
  Arms: Placebo group

SUMMARY:
The objective of this research is to assess the efficacy of oral metformin in mitigating the aging process in middle-aged and elderly males, to pinpoint sensitive indicators of human senescence, and to offer innovative frameworks and scientific insights for pharmaceutical interventions in aging.

DETAILED DESCRIPTION:
Subjects in both the metformin hydrochloride extended-release tablets treatment group and the placebo group received two tablets (500 mg each) once daily after dinner, continuing for a one-year period of drug intervention.

ELIGIBILITY:
Inclusion Criteria：

1. Male
2. Age 55-65; 18-28;
3. Able to understand and execute instructions;
4. After reading the consent form, be able to answer questions about the study and demonstrate understanding of the protocol;
5. Be able to participate in regular follow-up visits.

Exclusion Criteria

1. Severe chronic or acute disease: cancer, clinically significant congestive heart failure, chronic obstructive pulmonary disease (COPD), previous or new-onset diabetes, inflammatory state, serum creatinine >1.5 mg/dl , active liver disease, History of metabolic acidosis, poorly controlled hypertension, epilepsy, recent (within 3 months) cardiovascular events (MI, PTCA, CABG, stroke), severe renal insufficiency, inflammatory bowel disease, persistent glucocorticoids Treatment; neurological diseases such as dementia, AD, PD, etc.; infectious diseases such as HIV, hepatitis, tuberculosis, etc.; severe autoimmune diseases;
2. BMI<18.5 or BMI>30;
3. Persistent alcohol or drug abuse;
4. Treatment with drugs known to affect glucose metabolism (other diabetes drugs, systemic glucocorticoids, niacin);
5. Hypersensitivity to metformin or any component of the preparation;
6. Have taken metformin, low-dose aspirin, acarbose, vitamin C in the recent (3 months);
7. Unable to provide informed consent;
8. Other circumstances in which the researcher believes that the physical factors of the participants may adversely affect the research process or results.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 130 (Estimated)
Dates: Start 2024-06-30 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Composite the efficacy of metformin in intervening aging | Baseline - 12 month
  1. Metformin delay aging related sensitive indicators (2), such as SA*, ancient virus *.
  2. Metformin inhibits markers of inflammation in the body (4), such as C1 protein *, CRP, CXCL9, TNFa.
  3. Metformin improved immune cell-related indicators (10*), such as T1/T2/L gene expression.
  4. Metformin improves metabolism-related indexes (4), such as metabolic secretion factors APOX1* and APOX2*.
  5. Age-related indicators have been published (5), such as telomere length, DNA methylation age, hormone levels, etc.

SECONDARY OUTCOMES:
Composite Through clinical physical examination data, behavioral indicators and multilevel omics data, to discover new sensitive biomarkers for evaluating aging. | Baseline - 12 month
  1. Aging atlas-R, PBMC RNA profiling, >5% DEGs.
  2. Aging atlas-P, proteomic profiling, >5% DEPs.
  3. Aging atlas-M, metabolic profiling, >5% metabolites.
  4. Aging atlas-B, metagenomic profiling, >5% microbiotas.
  5. Reduce human biological age complex parameters.

CONTACTS AND LOCATIONS:
Overall Officials: Guoguang Zhao, professor, Study Chair — Xuanwu Hospital, Beijing; Guoguang Zhao, professor, Principal Investigator — Xuanwu Hospital, Beijing; Jing Li, professor, Study Director — Xuanwu Hospital, Beijing
Locations (1):
- Xuanwu Hospital Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] de Villartay JP, Rouger P, Muller JY, Salmon C. HLA antigens on peripheral red blood cells: analysis by flow cytofluorometry using monoclonal antibodies. Tissue Antigens. 1985 Jul;26(1):12-9. doi: 10.1111/j.1399-0039.1985.tb00929.x. PMID 3898468
- [Background] Chai M, Jiang M, Vergnes L, Fu X, de Barros SC, Doan NB, Huang W, Chu J, Jiao J, Herschman H, Crooks GM, Reue K, Huang J. Stimulation of Hair Growth by Small Molecules that Activate Autophagy. Cell Rep. 2019 Jun 18;27(12):3413-3421.e3. doi: 10.1016/j.celrep.2019.05.070. PMID 31216464
- [Background] Foretz M, Guigas B, Bertrand L, Pollak M, Viollet B. Metformin: from mechanisms of action to therapies. Cell Metab. 2014 Dec 2;20(6):953-66. doi: 10.1016/j.cmet.2014.09.018. Epub 2014 Oct 30. PMID 25456737
- [Background] Garber AJ, Duncan TG, Goodman AM, Mills DJ, Rohlf JL. Efficacy of metformin in type II diabetes: results of a double-blind, placebo-controlled, dose-response trial. Am J Med. 1997 Dec;103(6):491-7. doi: 10.1016/s0002-9343(97)00254-4. PMID 9428832
- [Background] TODAY Study Group; Zeitler P, Hirst K, Pyle L, Linder B, Copeland K, Arslanian S, Cuttler L, Nathan DM, Tollefsen S, Wilfley D, Kaufman F. A clinical trial to maintain glycemic control in youth with type 2 diabetes. N Engl J Med. 2012 Jun 14;366(24):2247-56. doi: 10.1056/NEJMoa1109333. Epub 2012 Apr 29. PMID 22540912
- [Background] Cabreiro F, Au C, Leung KY, Vergara-Irigaray N, Cocheme HM, Noori T, Weinkove D, Schuster E, Greene ND, Gems D. Metformin retards aging in C. elegans by altering microbial folate and methionine metabolism. Cell. 2013 Mar 28;153(1):228-39. doi: 10.1016/j.cell.2013.02.035. PMID 23540700
- [Background] Gronich N, Rennert G. Beyond aspirin-cancer prevention with statins, metformin and bisphosphonates. Nat Rev Clin Oncol. 2013 Nov;10(11):625-42. doi: 10.1038/nrclinonc.2013.169. Epub 2013 Oct 1. PMID 24080598
- [Background] Kodali M, Attaluri S, Madhu LN, Shuai B, Upadhya R, Gonzalez JJ, Rao X, Shetty AK. Metformin treatment in late middle age improves cognitive function with alleviation of microglial activation and enhancement of autophagy in the hippocampus. Aging Cell. 2021 Feb;20(2):e13277. doi: 10.1111/acel.13277. Epub 2021 Jan 14. PMID 33443781
- [Background] Kulkarni AS, Gubbi S, Barzilai N. Benefits of Metformin in Attenuating the Hallmarks of Aging. Cell Metab. 2020 Jul 7;32(1):15-30. doi: 10.1016/j.cmet.2020.04.001. Epub 2020 Apr 24. PMID 32333835
- [Background] Li C, Mu N, Gu C, Liu M, Yang Z, Yin Y, Chen M, Wang Y, Han Y, Yu L, Ma H. Metformin mediates cardioprotection against aging-induced ischemic necroptosis. Aging Cell. 2020 Feb;19(2):e13096. doi: 10.1111/acel.13096. Epub 2020 Jan 14. PMID 31944526
- [Background] Williams-Herman D, Johnson J, Teng R, Golm G, Kaufman KD, Goldstein BJ, Amatruda JM. Efficacy and safety of sitagliptin and metformin as initial combination therapy and as monotherapy over 2 years in patients with type 2 diabetes. Diabetes Obes Metab. 2010 May;12(5):442-51. doi: 10.1111/j.1463-1326.2010.01204.x. PMID 20415693
- [Background] Neumann B, Baror R, Zhao C, Segel M, Dietmann S, Rawji KS, Foerster S, McClain CR, Chalut K, van Wijngaarden P, Franklin RJM. Metformin Restores CNS Remyelination Capacity by Rejuvenating Aged Stem Cells. Cell Stem Cell. 2019 Oct 3;25(4):473-485.e8. doi: 10.1016/j.stem.2019.08.015. PMID 31585093
- [Background] Martin-Montalvo A, Mercken EM, Mitchell SJ, Palacios HH, Mote PL, Scheibye-Knudsen M, Gomes AP, Ward TM, Minor RK, Blouin MJ, Schwab M, Pollak M, Zhang Y, Yu Y, Becker KG, Bohr VA, Ingram DK, Sinclair DA, Wolf NS, Spindler SR, Bernier M, de Cabo R. Metformin improves healthspan and lifespan in mice. Nat Commun. 2013;4:2192. doi: 10.1038/ncomms3192. PMID 23900241
- [Background] Ma T, Tian X, Zhang B, Li M, Wang Y, Yang C, Wu J, Wei X, Qu Q, Yu Y, Long S, Feng JW, Li C, Zhang C, Xie C, Wu Y, Xu Z, Chen J, Yu Y, Huang X, He Y, Yao L, Zhang L, Zhu M, Wang W, Wang ZC, Zhang M, Bao Y, Jia W, Lin SY, Ye Z, Piao HL, Deng X, Zhang CS, Lin SC. Low-dose metformin targets the lysosomal AMPK pathway through PEN2. Nature. 2022 Mar;603(7899):159-165. doi: 10.1038/s41586-022-04431-8. Epub 2022 Feb 23. PMID 35197629
- [Background] Lopez-Otin C, Blasco MA, Partridge L, Serrano M, Kroemer G. Hallmarks of aging: An expanding universe. Cell. 2023 Jan 19;186(2):243-278. doi: 10.1016/j.cell.2022.11.001. Epub 2023 Jan 3. PMID 36599349